CLINICAL TRIAL: NCT04483011
Title: A Randomized, Double-blind, Comparator-controlled, Cross-over Study to Investigate the Safety and Efficacy of RiaGev™ in Healthy Adults
Brief Title: The Safety and Efficacy Study of RiaGev in Healthy Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bioenergy Life Science, Inc. (Industry)
Collaborators: KGK Science Inc. (Industry); University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 19RNHB(1918)
Record Dates: First submitted 2020-06-24; First posted 2020-07-23 (Actual); Results first posted 2020-11-25 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Metabolic Syndrome; Premature Aging
Keywords: NAD+; ATP; Glutathione; Cortisol; Exercise
MeSH Terms: conditions — Metabolic Syndrome; Aging, Premature; Motor Activity

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, comparator-controlled, cross-over
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RiaGev (Experimental): RiaGev, 2000mg, BID
  Interventions: Dietary Supplement: RiaGev
- Comparator (Active Comparator): Comparator matched to RiaGev, BID
  Interventions: Dietary Supplement: RiaGev

INTERVENTIONS:
Dietary Supplement: RiaGev — Dietary supplementation

SUMMARY:
This current randomized, double-blind, comparator-controlled, cross over study investigates the efficacy and safety of RiaGev™ via evaluation of NAD+, ATP, glucose, insulin, glutathione, and cortisol levels in healthy adults of ages 36-65.

DETAILED DESCRIPTION:
Nicotinamide adenine dinucleotide (NAD+) is one of the essential cofactors required for the proper function of living cells, and depletion in NAD has been correlated to aging individuals as NAD is associated with oxidative stress and energy production. Per the Population Reference Bureau (PRB), it is estimated that by the year 2060, the number of Americans over the age of 65 will double to over 98 million. As well, over the years, there has been a continuous rise in obesity within older Americans, reaching 44% for women and 36% for men in the age range of 65-74. One of the most common chronic diseases that are accompanied by aging and obesity diabetes. In 2016 the WHO reported that approximately 1.6 million deaths were attributed to diabetes. Half of these individuals had high blood glucose before the age of 70. Hence it is crucial to actively control blood glucose and oxidative stress during one's midlife stage.

The investigating product RiaGev™ is the first and only commercially available product that contains Bioenergy Ribose® and vitamin B3. It increases NAD+ in the body efficiently to promote healthy mitochondria, active immunity, and cholesterol reduction. As a result, D-ribose is essential for healthy aging.

Bioenergy Ribose® is a 5-carbon carbohydrate (C5H10O5) called D-ribose designated as a Generally Recognized as Safe (GRAS) substance by the US Food and Drug Administration (FDA). It is produced via the pentose phosphate pathway (PPP), which is fundamental for adenosine triphosphate (ATP) production. The PPP is a rate-limiting step that makes use of a short supply enzyme called glucose-6-phosphate dehydrogenase (G-6-PDH). Supplementation of D-ribose can bypass the PPP and directly contribute to ATP production. In addition, to its function for ATP production D-ribose is a critical element of deoxyribonucleic acid (DNA), ribonucleic acid (RNA), and acetyl coenzyme A. Provided there is a reduction in ATP production; aging is frequently due to a decline in mitochondria function. Hence, cell function and integrity are compromised, leading to chronic cardiovascular conditions and fatigue (6). With active D-ribose supplementation, improvements have been noted in several pathological conditions such as chronic fatigue syndrome, fibromyalgia, and myocardial dysfunction. Furthermore, D-ribose demonstrated improvements in athletic performances by recovering ATP levels and repairing cellular damage.

Vitamin B3 is an essential water-soluble vitamin known as either niacin, nicotinic acid, or nicotinamide. It is found in foods such as chicken, beef, fish, nuts, legumes, and grains. Also, vitamin B3 can be obtained from conversions of tryptophan in the body. Therefore, foods with tryptophan such as milk, eggs, meat, and fish are another great source of vitamin B3. Once vitamin B3 is consumed, it is converted into two different active forms called NAD+ or nicotinamide adenine dinucleotide phosphate (NADP). NAD+ and NADP are essential for various metabolic redox processes with oxidized or reduced substrates. Cellular functions like genome integrity, gene expression, and cellular communication are carried out by NAD+ required enzymes. These required enzymes are also crucial for the production of ATP via energy transfer from carbohydrates, fats, and proteins. NADP is involved in fewer reactions than NAD+ such as cholesterol and fatty acid synthesis along with antioxidation. Lack of NAD+ has been associated with a variety of aging-related conditions such as metabolic syndrome, cardiovascular health, and cancer.

This current randomized, double-blind, comparator-controlled, cross over study will investigate the efficacy and safety of RiaGev™ via evaluation of NAD+, glucose, insulin, glutathione, and cortisol levels in healthy adults of ages 36-65.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and females between the ages of 35 and 65 years of age, inclusive
2. BMI between 18.5 to 29.9 kg/m2, inclusive
3. Female participant is not of child-bearing potential, defined as females who have undergone a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation, complete endometrial ablation) or have been post-menopausal (natural or surgically) for at least 1 year prior to screening

   Or,

   Females of child-bearing potential must have a negative urine pregnancy test at screening and baseline and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:
   * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   * Double-barrier method
   * Intrauterine devices
   * Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
   * Vasectomy of partner at least 6 months prior to screening
4. Healthy as determined by laboratory results, medical history, physical exam and EKG
5. Agrees to avoid supplementation with tryptophan and vitamin B3 or its derivatives (niacin, nicotinic acid, niacinamide) one week prior to randomization and during the study
6. Ability to complete maximal and submaximal exercise tests
7. Agrees to maintain current diet and activity level throughout the study
8. Agrees to comply to all study procedures
9. Has given voluntary, written, informed consent to participate in the study
10. Self-reported good sleeper at screening. Have a regular sleep cycle with a bedtime between the approximate hours of 9:00pm and 12:00am and regularly receive between 7-9 hours of sleep, and agrees to maintain this sleep schedule throughout the study.

Exclusion Criteria:

1. Women who are pregnant, breast feeding, or planning to become pregnant during the trial
2. Allergy or sensitivity to investigational product's ingredients or standard meal provided
3. Current or ex-smokers within the past year
4. Major surgery within the past 3 months which may impact the study outcomes to be assessed by the QI.
5. Untreated/unresolved/uncontrolled cardiovascular disease. Participants with no significant cardiovascular event in the past 1 year and on stable medication may be included after assessment by the QI on a case by case basis
6. Self reported current or pre-existing thyroid condition. Treatment on a stable dose medication for over 3 months will be reviewed on a case-by-case basis by the QI
7. Current or history of hypertension.
8. Type I or Type II diabetes
9. Cancer, except skin cancers completely excised with no chemotherapy or radiation with a follow up that is negative. Volunteers with cancer in full remission for more than five years after diagnosis are acceptable
10. Self reported of any autoimmune disease or immune-compromised
11. Self reported by subjects of being HIV or Hepatitis B/C positive
12. History or currently with kidney and liver diseases assessed by QI on a case by case basis, with the exception of history of kidney stones symptom free for 1 year
13. Known medical or psychological condition that, in the qualified investigator's opinion, could interfere with study participation
14. Significant gastrointestinal disease (examples include but are not limited to Celiac disease and inflammatory bowel disease)
15. Self reported of bleeding disorders.
16. Current diagnosis of gout within past three months as per the QI's assessment
17. Clinically significant abnormal laboratory results at screening as assessed by QI
18. Current use of prescribed medications or over the counter supplements that may interfere with the IP assessed by QI (See Section 7.3)
19. Alcohol consumption of >2 standard drinks/day or >14 drinks/week
20. Alcohol or drug abuse within the past 12 months
21. Use of medical marijuana
22. Frequent use of recreational drugs within 6 months of baseline assessed as per QI
23. Planned blood donation during or within 30 days following conclusion of clinical trial
24. Participation in other clinical research trials 30 days prior to baseline
25. Participants that are cognitively impaired and/or who are unable to give informed consent
26. Any other active or unstable medical condition, that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant.

Ages: 36 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-11-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Malkanthi Evans, Ph.D, Study Chair — KGK Science Inc.; Trisha Shamp, PA-C, Ph.D, Principal Investigator — Prism Research, Inc.
Locations (1):
- Prism Research, Inc., Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total of 42 subject screened, 18 enrolled into study and randomized into two groups with 9 subjects each.
Groups:
- RiaGev, Then Comparator: RiaGev, 2000mg, BID, in Intervention Period 1, then 7 day washout, then cross-over to Comparator in Intervention Period 2
- Comparator, Then RiaGev: Comparator, BID, in Intervention Period 1, then 7 day washout, then cross-over to RiaGev 2000mg BID in Intervention Period 2
Period: Intervention Period 1 (8 Days)
Arm/Group | RiaGev, Then Comparator | Comparator, Then RiaGev
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0
Period: Washout (7 Days)
Arm/Group | RiaGev, Then Comparator | Comparator, Then RiaGev
Started | 9 | 9
Completed | 9 | 8
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Intervention Period 2 (8 Days)
Arm/Group | RiaGev, Then Comparator | Comparator, Then RiaGev
Started | 9 | 8
Completed | 9 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- RiaGev, Then Comarator: RiaGev, 2000mg, BID, in Period 1, then cross-over to Comparator in Period 2, after 7-day washout.
- Comparator, Then RiaGev: Comparator, BID, in Period 1, then cross-over to RiaGev 2000mg, BID, in Period 2 after 7-day washout.
- Total: Total of all reporting groups
Arm/Group | RiaGev, Then Comarator | Comparator, Then RiaGev | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.11 (8.62) | 53.33 (7.31) | 51.72 (7.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 9 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18
Weight [Mean (Standard Deviation); unit: Kg] | 75.15 (14.60) | 79.06 (19.99) | 77.11 (17.30)
Height [Mean (Standard Deviation); unit: CM] | 175.22 (8.12) | 172.67 (14.18) | 173.95 (11.09)
BMI [Mean (Standard Deviation); unit: Kg/cm^2] | 24.29 (2.96) | 26.12 (2.75) | 25.21 (2.86)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 124.57 (13.01) | 124.26 (9.32) | 124.42 (11.16)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 78.33 (7.63) | 78.31 (5.01) | 78.32 (6.32)
Heart Rate [Mean (Standard Deviation); unit: bpm] | 64.11 (19.62) | 66.33 (9.11) | 65.22 (14.35)

OUTCOME MEASURES:

1. Primary Outcome: Whole Blood NAD+ Level Change Over Baseline After Supplementation
Description: Whole blood NAD+ concentration are measured at Day 1, Day 3, Day 5, and Day 8. A NAD+ Level change over baseline (Day 1) is calculated by subtracting the NAD+ level at Day 1 ( e.g Day 5 over Day 1 = Day 5 - Day 1). The significance of change (p value) is calculated comparing within RiaGev or Comparator group, and between RiaGev and Comparator groups.
Time Frame: Day 1 to Day 8
Population: ITT
Measure: Mean (Standard Deviation); unit: MicroMolar
Groups:
- Comparator: Comparator matched to RiaGev, BID
  Comparator: Dietary ingredients
Arm/Group | RiaGev | Comparator
Number analyzed (Participants) | 18 | 17
MicroMolar
  Day 3 over Day 1 | 1.23 (3.39) | 0.13 (4.83)
  Day 5 over Day 1 | 2.12 (4.72) | -0.20 (2.79)
  Day 8 over Day 1 | 1.30 (3.20) | -0.60 (2.53)
Statistical Analysis 1: Comparison: RiaGev; A comparison between before and after RiaGev supplementation; Test type: Superiority; p = 0.034, Wilcoxon (Mann-Whitney) — < 0.05; Mean Difference (Net) = 2.12, Standard Deviation 4.72 — The p value in RiaGev group at Day 5 over Dave 1 is reported
Statistical Analysis 2: Comparison: Comparator; A comparison between before and after supplementation of Comparator; Test type: Superiority; p = 0.265, Wilcoxon (Mann-Whitney) — p > 0.05; Mean Difference (Net) = -0.20, Standard Deviation 2.79 — The p value in Comparator group at Day 5 over Day 1 is reported
Statistical Analysis 3: Comparison: RiaGev vs Comparator; A comparison between RiaGev and Comparator groups; Test type: Superiority; p = 0.044, ANCOVA — < 0.05; Mean Difference (Net) = 2.12, Standard Deviation 4.72 — The p value between RiaGev and Comparator groups at Day 5 over Day 1 is reported

2. Primary Outcome: Whole Blood NADP+ Level Change Over Baseline After Supplementation
Description: Whole blood NADP+ concentration are measured at Day 1, Day 3, Day 5, and Day 8. NADP+ level changes over baseline (Day 1) are calculated by substracting NADP+ level at Day 1. The significance of change (p values) are calculated comparing changes within and between RiaGev and Comparator groups.
Time Frame: Day 1 to Day 8
Population: ITT
Measure: Mean (Standard Deviation); unit: microMolar
Arm/Group | RiaGev | Comparator
Number analyzed (Participants) | 18 | 17
microMolar
  Day 3 over Day 1 | 1.30 (1.72) | 0.85 (2.49)
  Day 5 over Day 1 | 1.88 (2.55) | 0.51 (1.52)
  Day 8 over Day 1 | 1.33 (1.88) | 0.34 (1.34)
Statistical Analysis 1: Comparison: RiaGev; A comparison between before and after supplementation of RiaGev; Test type: Superiority; p = 0.008, Wilcoxon (Mann-Whitney) — p < 0.05; Mean Difference (Net) = 1.33, Standard Deviation 1.88 — The p value in RiaGev group at Day 5 over Day 1 is reported
Statistical Analysis 2: Comparison: Comparator; A comparison between before and after supplementation with Comparator; Test type: Superiority; p = 0.297, Wilcoxon (Mann-Whitney) — p > 0.05; Mean Difference (Net) = 0.34, Standard Deviation 1.34 — The p value in Comparator group at Day 5 over Day 1 is reported
Statistical Analysis 3: Comparison: RiaGev vs Comparator; A comparison between RiaGev and Comparator supplementation; Test type: Superiority; p = 0.04, ANCOVA — p < 0.05; Mean Difference (Net) = 1.33, Standard Deviation 1.88 — The p value between RiaGev and Comparator groups at Day 5 over Day 1 is reported

3. Primary Outcome: Whole Blood NAD+ Plus NADP+ Level Change Over Baseline
Description: The change in whole blood NAD+ plus NADP+ levels from Day 1 baseline to Day 8 when supplemented with RiaGev™ or comparator. The parameter is measured at Day 1, Day 3, Day 5, and Day 8. A change over baseline is calculated by subtracting Day 1 value. The significance of changes (p value) are calculated by comparing within and between RiaGev and Comparator groups.
Time Frame: Day 1 to 8
Population: ITT population
Measure: Mean (Standard Deviation); unit: microMolar
Groups:
- Comparator: Comparator matched to RiaGev, BID
  Comparator: Dietary ingredient
Arm/Group | RiaGev | Comparator
Number analyzed (Participants) | 18 | 17
microMolar
  Day 3 over Day 1 | 2.54 (4.60) | 0.97 (7.10)
  Day 5 over Day 1 | 4.01 (6.57) | 0.40 (3.88)
  Day 8 over Day 1 | 2.63 (4.30) | -0.24 (3.39)
Statistical Analysis 1: Comparison: RiaGev; A comparison between before and after RiaGev supplementation; Test type: Superiority; p = 0.004, Wilcoxon (Mann-Whitney) — p < 0.05; Mean Difference (Net) = 4.01, Standard Deviation 6.57 — The p value in the RiaGev group at Day 5 over Day 1 is reported
Statistical Analysis 2: Comparison: Comparator; A comparison between before and after supplementation with Comparator; Test type: Superiority; p = 0.640, Wilcoxon (Mann-Whitney) — p > 0.05; Mean Difference (Net) = 0.40, Standard Deviation 3.88 — The p value in Comparator group at Day 5 over Day 1 is reported
Statistical Analysis 3: Comparison: RiaGev vs Comparator; A comparison between RiaGev and Comparator supplementation; Test type: Superiority; p = 0.014, ANCOVA — p < 0.05; Mean Difference (Net) = 4.01, Standard Deviation 6.57 — The p value between RiaGev and Comparator groups at Day 5 over Day 1 is reported

4. Secondary Outcome: Serum Glucose Change After RiaGev Supplementation Assessed by OGTT
Description: The serum glucose as assessed by a standard Oral Glucose Tolerance Test (OGTT) on Day 1 and on Day 8 after 7-day supplementation with either RiaGev™ or comparator. Incremental Area Under the Curve (iAUC) is used as overall blood glucose. Serum glucose change is calculated by subtracting iAUC on Day 1 from iAUC on Day 8. The significance of change (p value) is calculated by comparing values on Day 8 and Day 1.
Time Frame: 7 days
Population: ITT population
Measure: Mean (Standard Deviation); unit: (mg/dL)*min
Arm/Group | RiaGev | Comparator
Number analyzed (Participants) | 18 | 17
(mg/dL)*min
  Day 1 | 17700.42 (2525.30) | 876.25 (1601.18)
  Day 8 | 662.50 (2031.70) | 574.17 (1640.77)
  Change from Day 1 to Day 8 | -1037.92 (1590.74) | -302.08 (1427.42)
Statistical Analysis 1: Comparison: RiaGev; A comparison before and after RiaGev supplementation; Test type: Superiority; p = 0.013, Wilcoxon (Mann-Whitney) — p < 0.05; Mean Difference (Net) = -1037.92, Standard Deviation 1590.74 — The p value in RiaGev group at Day 8 over Day 1 is reported
Statistical Analysis 2: Comparison: Comparator; A comparison before before and after supplementation with Comparator; Test type: Superiority; p = 0.382, Wilcoxon (Mann-Whitney) — p > 0.05; Mean Difference (Net) = -302.08, Standard Deviation 1427.42 — The p value in Comparator group at Day 8 over Day 1 is reported

5. Secondary Outcome: Serum Insulin Change After RiaGev Supplementation Assessed by OGTT
Description: Serum insulin is assessed by a standard Oral Glucose Tolerance Test (OGTT) on Day 1 and Day 8 after 7-day supplementation with either RiaGev™ or comparator. Serum insulin change is calculated by substracting its level on Day 1 from Day 8. The significance of change (p value) is calculated by comparing Day 1 and Day 8.
Time Frame: 7 days
Population: ITT population
Measure: Mean (Standard Deviation); unit: (microUnit/mL)*min
Arm/Group | RiaGev | Comparator
Number analyzed (Participants) | 18 | 17
(microUnit/mL)*min
  Day 1 | 4807.42 (2419.04) | 4545.67 (1915.67)
  Day 8 | 4672.29 (2427.27) | 4410.88 (1929.12)
  Change from Day 1 to Day 8 | -135.13 (2153.66) | -134.79 (1830.16)
Statistical Analysis 1: Comparison: RiaGev; A comparison between before and after RiaGev supplementation; Test type: Superiority; p = 0.793, Wilcoxon (Mann-Whitney) — p > 0.05; Mean Difference (Net) = -135.13, Standard Deviation 2153.66 — The p value in RiaGev group at Day 8 over Day 1 baseline is reported
Statistical Analysis 2: Comparison: Comparator; A comparison between before and after supplementation with Comparator; Test type: Superiority; p = 0.758, Wilcoxon (Mann-Whitney) — p > 0.05; Mean Difference (Net) = -134.79, Standard Deviation 1830.16 — The p value in Comparator group at Day 8 over Day 1 baseline is reported

6. Secondary Outcome: Serum Glutathione (GSH + GSSG) Change Over Baseline After RiaGev Supplementation
Description: Total serum Glutathione (GSH + GSSG) is measured on Day 1, Day 3, Day 5 and Day 8. after a 7-day supplementation with either RiaGev™ or comparator. A change over baseline is calculated by subtracting glutathione level on Day 1 baseline (e g Day 5 over Day 1 = Day 5 - Day 1). The significance of change (p value) is calculated within the RiaGev or Comparator group.
Time Frame: 7 days
Population: ITT
Measure: Mean (Standard Deviation); unit: microMolar
Arm/Group | RiaGev | Comparator
Number analyzed (Participants) | 18 | 17
microMolar
  Day 3 over Day 1 | 61.85 (124.73) | 32.43 (130.37)
  Day 5 over Day 1 | 70.20 (123.89) | 15.55 (88.62)
  Day 8 over Day 1 | 9.55 (66.82) | -15.08 (76.05)
Statistical Analysis 1: Comparison: RiaGev; A comparison between before and after RiaGev supplementation; Test type: Superiority; p = 0.003, Wilcoxon (Mann-Whitney) — p < 0.05; Mean Difference (Net) = 70.20, Standard Deviation 123.89 — The p value in RiaGev group at Day 5 over Day 1 is reported
Statistical Analysis 2: Comparison: Comparator; A comparison between before and after supplementation with Comparator; Test type: Superiority; p = 0.766, Wilcoxon (Mann-Whitney) — p > 0.05; Mean Difference (Net) = 15.55, Standard Deviation 88.62 — The p value in Comparator group at Day 5 over Day 1 is reported

7. Secondary Outcome: Serum High Energy Phosphate (ATP + ADP) Concentration After RiaGev Supplementation
Description: Serum high energy phosphate (ATP + ADP) after a 7-day supplementation with either RiaGev™ or comparator. The measurement take place on Day 1, Day 3, Day 5, and Day 8. Comparison are made between the two groups. The significance (p value) is also calculated between the groups.
Time Frame: 7 days
Population: ITT
Measure: Mean (Standard Deviation); unit: microMolar
Arm/Group | RiaGev | Comparator
Number analyzed (Participants) | 18 | 17
microMolar
  Day 1 (baseline) | 327.10 (42.87) | 324.94 (58.55)
  Day 3 | 351.18 (75.71) | 345.98 (102.56)
  Day 5 | 353.28 (82.03) | 329.27 (94.34)
  Day 8 | 330.40 (41.89) | 326.20 (45.46)
Statistical Analysis 1: Comparison: RiaGev vs Comparator; A comparison between RiaGev and Comparator groups after 7-day supplementation; Test type: Superiority; p = 0.029, ANCOVA — p < 0.05; Mean Difference (Net) = 24.01, Standard Deviation 58.20 — The p value between RiaGev and Comparator groups at Day 5 is reported

8. Secondary Outcome: The Waking Salivary Cortisol Level After RiaGev Supplementation
Description: The salivary cortisol level after a 7-day supplementation with either RiaGev™ or comparator. The measurement take place on Day 1, 3, 5, and 8. The salivary cortisol level as well as change of salivary cortisol level over baseline (Day 1) are reported. Comparisons are make both between the RiaGev and Comparison groups as well as within RiaGev group against its Day 1 baseline. The corresponding significance (p value) will be calculated.
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: mcg/dL
Arm/Group | RiaGev | Comparator
Number analyzed (Participants) | 18 | 17
mcg/dL
  Day 1 (baseline) | 0.43 (0.15) | 0.51 (0.24)
  Day 3 | 0.40 (0.19) | 0.47 (0.19)
  Day 5 | 0.41 (0.32) | 0.57 (0.29)
  Day 8 | 0.38 (0.18) | 0.51 (0.22)
  Day 3 over Day 1 | -0.03 (0.18) | -0.04 (0.26)
  Day 5 over Day 1 | -0.02 (0.34) | 0.07 (0.36)
  Day 8 over Day 1 | -0.05 (0.19) | 0.00 (0.28)
Statistical Analysis 1: Comparison: RiaGev vs Comparator; A comparison between RiaGev and Comparator groups; Test type: Superiority; p = 0.034, ANCOVA — p < 0.05; Mean Difference (Net) = -0.16, Standard Deviation 0.32 — The p value between RiaGev and Comparator groups at Day 5 is reported

9. Secondary Outcome: The Change in Checklist Individual Strength (CIS) Questionnaire Outcome After a 7-day Supplementation With Either RiaGev™ or Comparator.
Description: Checklist Individual Strength (CIS) Questionnaire was designed by the Dutch research team of Vercoulen et el, to measure fatigues. A standard CIS Questionnaire contains 20 questions, each scoring 1 to 7, total score 20 - 140, with higher score indicating more tiredness. Thus, a negative value in changing score (such as Day 5 - Day 1 baseline) means reduction of tiredness and verse versa.
Time Frame: 7 days
Population: ITT
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | RiaGev | Comparator
Number analyzed (Participants) | 18 | 17
Score on a scale
  Day 3 over Day 1 | -9.78 (13.45) | -4.28 (5.93)
  Day 5 over Day 1 | -8.33 (12.99) | -2.56 (5.66)
  Day 8 over Day 1 | -5.78 (16.27) | -1.67 (7.54)
Statistical Analysis 1: Comparison: RiaGev; A comparison between before and after RiaGev supplementation; Test type: Superiority; p = 0.014, Wilcoxon (Mann-Whitney) — p < 0.05; Mean Difference (Net) = -8.33, Standard Deviation 12.99 — The p value in RiaGev group at Day 5 over Day 1 is reported
Statistical Analysis 2: Comparison: Comparator; A comparison between before and after supplementation with Comparator; Test type: Superiority; p = 0.049, Wilcoxon (Mann-Whitney) — p < 0.05; Mean Difference (Net) = -2.56, Standard Deviation 5.66 — The p value in Comparator group at Day 5 over Day 1 is reported

10. Other Pre Specified Outcome: The Number of Out-of-norm Clinical Chemistry Parameters When Supplemented With RiaGev or Comparator
Description: The number of out-of-norm incidence (as indicator of safety) will be reported. Clinical chemistry parameters including alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin, creatinine, electrolytes (Na, K, Cl), fasting glucose. When a parameter is within normal limit, it will been reported as 0 out-of-norm.
Time Frame: 7 days
Population: ITT Populaiton
Measure: Count of Participants; unit: Participants
Arm/Group | RiaGev | Comparator
Number analyzed (Participants) | 18 | 17
Participants
  Creatine Clearance | 0 | 0
  Creatinine | 0 | 0
  Fasting Blood Glucose | 0 | 0
  Aspartate Transaminase (AST) | 0 | 0
  Alanine Transaminase (ALT) | 0 | 0
  Chloride | 0 | 0
  Potassium | 0 | 0
  Sodium | 0 | 0
  Bilirubin | 0 | 0
  Hemoglobin A1c | 0 | 0
  Estimated Average Glucose | 0 | 0

11. Other Pre Specified Outcome: The Number of Out-of-norm Hematology Parameters When Supplemented With RiaGev or Comparator.
Description: The number of out-of-norm hematology parameter incidence (as indicator of safety) will be reported. Hematology parameters include white blood cell (WBC) count with differential (neutrophils, lymphocytes, monocytes, eosinophils, basophils), red blood cell (RBC) count, hemoglobin, hematocrit, platelet count, RBC indices (mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), red cell distribution width (RDW). When a parameter is within normal limits, it is reported as 0 out-of-norm.
Time Frame: 7 days
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | RiaGev | Comparator
Number analyzed (Participants) | 18 | 17
Participants
  White Blood Cell Counts | 0 | 0
  Red Blood Cell Counts | 0 | 0
  Hemoglobin | 0 | 0
  Hemotocrit | 0 | 0
  Mean Corpuscular Volume | 0 | 0
  Mean Corpuscular Hemoglobin | 0 | 0
  Mean Corpuscular Hemoglobin Concentration | 0 | 0
  Red Blood Cell Distribution Width | 0 | 0
  Platelet | 0 | 0
  Meran Package Volume | 0 | 0
  Nucleated Red Blood Cells (NRBCA) | 0 | 0
  Instrument Absolute Neotrophil Count (IANC) | 0 | 0
  Immature Granulocytes (IGAB) | 0 | 0
  Absolute Neutrophil Counts | 0 | 0
  Absolute Lymphocyte Count | 0 | 0
  Absolute Monocyte Count | 0 | 0
  Absolute Eosinophil Counts | 0 | 0
  Absolute Basophil Count | 0 | 0

12. Other Pre Specified Outcome: The Number of Out-of-norm Vital Signs When Supplemented With RiaGev or Comparator
Description: Vital signs include blood pressure (BP) and heart rate (HR). The number of out-of-norm incidence will be reported. When a parameter is within normal limits, it is reported as 0 out-of-norm.
Time Frame: 7 days
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | RiaGev | Comparator
Number analyzed (Participants) | 18 | 17
Participants
  Systolic Pressure | 0 | 0
  Diastolic Pressure | 0 | 0
  Heart Rate | 0 | 0

ADVERSE EVENTS:
Time Frame: 22 days
Description: Total number of post-emergent adverse events that are possibly relevant to the study.
Arm/Group | RiaGev | Comparator
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 1/18 | 1/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RiaGev (N=18) | Comparator (N=17)
Asthenia (General disorders) | 1 (1) | 0 (0) — Weakness, Resolved.
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Anorexia, Resolved.
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Joint Pain, Resolved

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2020-06-24): https://cdn.clinicaltrials.gov/large-docs/11/NCT04483011/SAP_000.pdf
  • Study Protocol (2019-10-07): https://cdn.clinicaltrials.gov/large-docs/11/NCT04483011/Prot_001.pdf